CLINICAL TRIAL: NCT03707366
Title: Fostering Healthy Futures for Teens: A Randomized Controlled Trial
Brief Title: Fostering Healthy Futures for Teens: An RCT
Acronym: FHF-T
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Denver (Other)
Responsible Party: Principal Investigator, Heather Taussig, Professor and Associate Dean for Research, University of Denver
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DU FHF-T
Record Dates: First submitted 2017-05-23; First posted 2018-10-16 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Child Abuse; Child Neglect; Risk Behavior; Delinquency; Mental Health Impairment; Substance Use; Educational Problems; Adolescent Development; Adolescent Behavior; Sexual Behavior; Child Maltreatment
Keywords: Mentoring; Positive Youth Development; Skills training; Relationships; Child Welfare
MeSH Terms: conditions — Risk-Taking; Substance-Related Disorders; Adolescent Behavior; Sexual Behavior

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with 2 groups
Who Masked: Outcomes Assessor
Masking Description: Research assistants who conduct the interviews are masked to condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FHF-T Intervention Group (Experimental): 9 months of 1:1 youth mentoring by graduate-student mentors; workshops; educational advocacy
  Interventions: Behavioral: FHF-T
- Control group (No Intervention): Services as usual

INTERVENTIONS:
Behavioral: FHF-T — FHF-T employs mentoring, consisting of relationship development, advocating for and empowering youth, and skill-building activities to promote positive youth development. Mentors meet individually for 2-3 hours per week for 30 weeks with each teen they mentor, in order to engage teens in positive youth development activities and provide skills training in areas including emotion recognition, perspective-taking, problem solving, effective communication, managing anger, healthy coping and resisting peer pressure for deviant activities. Youth also attend group workshops over the course of the program, in which they engage with other participants and mentors in skill-building activities.
  Arms: FHF-T Intervention Group

SUMMARY:
This study will implement and evaluate a mentoring program designed to promote positive youth development and reduce adverse outcomes among maltreated adolescents with open child welfare cases. Teenagers who have been maltreated are at heightened risk for involvement in delinquency, substance use, and educational failure as a result of disrupted attachments with caregivers and exposure to violence within their homes and communities. Although youth mentoring is a widely used prevention approach nationally, it has not been rigorously studied for its effects in preventing these adverse outcomes among maltreated youth involved in the child welfare system. This randomized controlled trial will permit us to implement and evaluate the Fostering Healthy Futures for Teens (FHF-T) program, which will use mentoring and skills training within an innovative positive youth development (PYD) framework to promote adaptive functioning and prevent adverse outcomes. Graduate student mentors will deliver 9 months of prevention programming in teenagers' homes and communities. Mentors will focus on helping youth set and reach goals that will improve their functioning in five targeted "REACH" domains: Relationships, Education, Activities, Career, and Health. In reaching those goals, mentors will help youth build social-emotional skills associated with preventing adverse outcomes (e.g., emotion regulation, communication, problem solving). The randomized controlled trial will enroll 234 racially and ethnically diverse 8th and 9th grade youth (117 intervention, 117 control), who will provide data at baseline prior to randomization, immediately post-program and 15 months post program follow-up. The aims of the study include testing the efficacy of FHF-T for high-risk 8th and 9th graders in preventing adverse outcomes and examining whether better functioning in positive youth development domains mediates intervention effects. It is hypothesized that youth randomly assigned to the FHF-T prevention condition, relative to youth assigned to the control condition, will evidence better functioning on indices of positive youth development in the REACH domains leading to better long-term outcomes, including adaptive functioning, high school graduation, career attainment/employment, healthy relationships, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Teens with open child welfare cases placed in foster care, kinship care or living at home
* Starting 8th or 9th grade
* History of child maltreatment according to child welfare and court records
* Live within 35 minutes of the University of Denver (for mentoring feasibility)

Exclusion Criteria:

* Youth with a known history of severe violent behavior and/or sexual perpetration
* Youth who are deemed unsafe or unable to participate in a community-based mentoring program by their caseworker
* Incarcerated at baseline
* Moderate or severe developmental delay or physical disability
* Youth who are/will be parenting during the prevention program

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 234 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Court filings for delinquency immediately post intervention | immediately post-intervention (T2)
  Presence of a court filing in administrative records for delinquent behavior
Court filings for delinquency 15 months-post intervention | 15-months-post intervention (T3)
  Presence of a court filing in administrative records for delinquent behavior
Self-reported delinquency immediately post intervention | immediately post-intervention (T2)
  The Adolescent Risk Behavior Survey (ARBS), a youth-report measure that assesses engagement in risk behaviors, will assess any delinquency, number of types of delinquency, any violent delinquency, and any non-violent delinquency
Self-reported delinquency 15 months-post intervention | 15-months-post intervention (T3)
  The Adolescent Risk Behavior Survey (ARBS), a youth-report measure that assesses engagement in risk behaviors, will assess any delinquency, number of types of delinquency, any violent delinquency, and any non-violent delinquency
School suspensions immediately post intervention | immediately post-intervention (T2)
  Any youth reported school suspensions, assessed by the Adolescent Risk Behavior Survey (ARBS), a youth-report measure that assesses engagement in risk behaviors
School suspensions 15 months-post intervention | 15-months-post intervention (T3)
  Any youth reported school suspensions, assessed by the Adolescent Risk Behavior Survey (ARBS), a youth-report measure that assesses engagement in risk behaviors
Substance use immediately post intervention | immediately post-intervention (T2)
  Self-reported number of types and frequency of substance use as assessed by the substance use scale of the Adolescent Risk Behavior Survey (ARBS), a youth-report measure that assesses engagement in risk behaviors
Substance use 15 months-post intervention | 15-months-post intervention (T3)
  Self-reported number of types and frequency of substance use as assessed by the substance use scale of the Adolescent Risk Behavior Survey (ARBS), a youth-report measure that assesses engagement in risk behaviors
Passing grades immediately post intervention | immediately post-intervention (T2)
  Youth report of passing all core academic courses, as assessed via researcher developed educational measure
Passing grades 15 months-post intervention | 15-months-post intervention (T3)
  Youth report of passing all core academic courses, as assessed via researcher developed educational measure

SECONDARY OUTCOMES:
Quality of Life | Baseline (T1), immediately post-intervention (T2) and 15-months-post intervention (T3)
  Self-reported mean quality of life as measured by the Life Satisfaction Scale (Andrews & Withey, 1976)
Extracurricular activity involvement | Baseline (T1), immediately post-intervention (T2) and 15-months-post intervention (T3)
  Self-reported number and frequency of extracurricular activity involvement will be measured by The Activities Scale, a project-designed measure.
Connectedness to school | Baseline (T1), immediately post-intervention (T2) and 15-months-post intervention (T3)
  Self-reported school connection will be measured by the mean score on the Psychological Sense of School Membership Scale (Goodenow, 1993) which assesses attachment and emotional response to a school environment.
Academic achievement | Baseline (T1), immediately post-intervention (T2) and 15-months-post intervention (T3)
  Academic Achievement will be assessed using standard scores on The Wechsler Individual Achievement Test Screener (WIAT Screener; Psychological Corporation, 1992).
Perceived Opportunities | Baseline (T1), immediately post-intervention (T2) and 15-months-post intervention (T3)
  Self-reported perceived opportunities will be assessed using mean scores on the Perceived Opportunities scale of the Adolescent Risk Behavior Survey (ARBS), a youth-report measure that assesses engagement in risk behaviors
Trauma symptoms | Baseline (T1), immediately post-intervention (T2) and 15-months-post intervention (T3)
  Self-reported trauma symptoms will be assessed using mean total and subscale scores of the Trauma Symptom Checklist (TSC; Briere, 1996).
Internalizing symptoms | Baseline (T1), immediately post-intervention (T2) and 15-months-post intervention (T3)
  Self-reported internalizing symptoms will be assessed using the mean score on the internalizing subscale of The Youth Self Report (YSR; Achenbach, 2001).
Externalizing symptoms | Baseline (T1), immediately post-intervention (T2) and 15-months-post intervention (T3)
  Self-reported externalizing symptoms will be assessed using the mean score on the externalizing subscale of The Youth Self Report (YSR; Achenbach, 2001).
Dating violence | Baseline (T1), immediately post-intervention (T2) and 15-months-post intervention (T3)
  Self-reported dating violence will be measured by The Conflict in Adolescent Dating Relationships Inventory (CADRI; Wolfe, Scott, Wekerle, & Pittman, 2001).
Coping skills | Baseline (T1), immediately post-intervention (T2) and 15-months-post intervention (T3)
  Self-reported coping skills will be measured using the mean scores on the subscales of the Children's Coping Strategies Checklist (Program for Prevention Research, 1999).
Conflict management skills | Baseline (T1), immediately post-intervention (T2) and 15-months-post intervention (T3)
  Self-reported conflict management skills will be measured using the mean score on the conflict management subscale of the Safe Dates Evaluation Questionnaire (Foshee, Bauman, Bennett, Suchindran, Benefield, & Linder, 2005).
Self-efficacy | Baseline (T1), immediately post-intervention (T2) and 15-months-post intervention (T3)
  Self-reported self-efficacy will be measured by the mean score on the Perceived Self-Efficacy Scale (Cowen, Work, Hightower, Wyman, Parker, & Ltyczewski, 1991).
Resiliency | Baseline (T1), immediately post-intervention (T2) and 15-months-post intervention (T3)
  Self-reported resiliency will be measured using standardized scores on The Resiliency Scales for Children and Adolescents (RSCA; Prince-Embury, 2006, 2007).
Help seeking behaviors | Baseline (T1), immediately post-intervention (T2) and 15-months-post intervention (T3)
  Self-reported help seeking will be measured by the number of identified social network members from whom the youth seek help and the frequency of seeking help on The Help Seeking Behaviors Scale (Pham, Y. K., McWhirter, E. H., & Murray, C., 2014).
Use of protection while having sex | Baseline (T1), immediately post-intervention (T2) and 15-months-post intervention (T3)
  Self-report of using protection while having sex, assessed by the Adolescent Risk Behavior Survey (ARBS), a youth-report measure that assesses engagement in risk behaviors

CONTACTS AND LOCATIONS:
Overall Officials: Heather Taussig, PhD, Principal Investigator — University of Denver; Kimberly Bender, PhD, Principal Investigator — University of Denver
Locations (1):
- University of Denver, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, Analytic Code

REFERENCES:
- [Background] Taussig H, Weiler L, Rhodes T, Hambrick E, Wertheimer R, Fireman O, Combs M. Fostering Healthy Futures for Teens: Adaptation of an Evidence-Based Program. J Soc Social Work Res. 2015 Dec;6(4):617-642. doi: 10.1086/684021. PMID 27019678
- [Result] Taussig, H.N., Bender, K., Bennett, R. Massey Combs, K., Fireman, O, & Wertheimer, R. (2020). Mentoring for teens with child welfare involvement: Permanency outcomes from a randomized controlled trial of the Fostering Healthy Futures for Teens program. Child Welfare, 97(5), 1-24.
- [Result] Taussig, H., Bender, K., Racz, S. & Evidence Based Policy Team, A. V. (2022, April 7). Fostering Healthy Futures for Teens. Retrieved from osf.io/673eu.
- Available data/document: Individual Participant Data Set — https://osf.io/673eu/